CLINICAL TRIAL: NCT01786174
Title: Phase IIa Double-Blind, Placebo-Controlled Study to Evaluate the Safety of Oral Fingolimod in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Gilenya in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ALS Therapy Development Institute (Other)
Responsible Party: Principal Investigator, James D. Berry MD, MGH Assistant Neurologist, HMS Instructor in Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P000313
Record Dates: First submitted 2013-02-04; First posted 2013-02-07 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Gilenya; Fingolimod
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gilenya (fingolimod) (Experimental): 0.5mg Gilenya (fingolimod) orally once daily for 28 days +/- 3 days
  Interventions: Drug: Gilenya
- Placebo (Placebo Comparator): 0.5mg placebo (sugar pill) orally once daily for 28 days +/- 3 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gilenya — 0.5mg Gilenya orally by mouth once daily for approximately 28 days
  Other Names: fingolimod
  Arms: Gilenya (fingolimod)
Other: Placebo — 0.5mg placebo (sugar pill) orally by mouth once daily for approximately 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Gilenya, also known as fingolimod, is safe and tolerable in patients with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
The primary objective of the study is to determine the acute safety and tolerability of oral administration of Gilenya (fingolimod) 0.5mg daily vs. matched oral placebo administered daily.

The primary outcome measure will be safety and tolerability; safety will be assessed by the occurrence of adverse events and clinically meaningful changes in vital signs, ophthalmologic examination, physical examination, electrocardiogram and standard clinical laboratory blood tests, and tolerability will be defined as the ability of subjects to complete the entire 4-week study.

The secondary outcome measure will be the measured effect of the treatment on circulating lymphocyte populations in patients with ALS.

Exploratory outcome measures will include the rate of decline of the ALS Functional Rating Scale (Revised) (ALSFRS-R) and Slow Vital Capacity (VC) during the course of treatment.

This study will be conducted in subjects who meet the El Escorial criteria of possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS. At screening, eligible subjects must be at least 18 years old, must have an SVC ≥ 65% of predicted capacity for age, height and gender, and must provide written informed consent prior to screening. Subjects on a stable dose of riluzole and those not taking riluzole, and women of child-bearing age at screening are eligible for inclusion as long as they meet specific protocol requirements.

Subjects will remain on randomized, placebo-controlled, double-blind treatment until the Week 4 visit. Each randomized subject will also have a Week 8 Follow-up Telephone Interview to assess for adverse events (AEs), changes in concomitant medications and to administer the ALSFRS-R.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria (Appendix 1).
3. Onset of weakness or spasticity due to ALS ≤ 2 years (24 months) prior to Baseline Visit.
4. Slow vital capacity (SVC) measure ≥65% of predicted for gender, height, and age at the screening visit.
5. Subjects must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days, prior to randomization (riluzole-naïve subjects are permitted in the study).
6. Subjects must be able to swallow oral medication at the Screening Visit and expected to be able to swallow the capsule throughout the course of the study.
7. Capable of providing informed consent and following trial procedures.
8. Geographically accessible to the site.
9. Women must not be able to become pregnant (e.g. post menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and three months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal (patch or contraceptive ring, for example) contraception), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.
10. Subjects must agree not to take live attenuated vaccines (including seasonal flu vaccine) 30 days before randomization, throughout the duration of the trial and for 60 days following the trial.

Exclusion Criteria:

1. Prior use of fingolimod (Gilenya®).
2. History or presence of cardiac conditions including:

   1. Cardiovascular or cerebrovascular disease in the previous 6 months (eg. myocardial infarction, unstable angina, or stroke)
   2. Congestive heart failure
   3. First, second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances
   4. Any history of Torsades de Pointes
3. Treatment with a prohibited medication within 30 days of the Baseline Visit:

   a. Class Ia or III antiarrhythmic medications: i.e., Quinidine, Sotalol Includes Nuedexta b. QT interval prolonging medications c. Ketoconazole d. Beta-blockers e. Calcium channel blockers f. Immunosuppressant medication g. Chemotherapeutic (anti-neoplastic) medications
4. Evidence on examination or ECG of bradycardia (<55 bpm), QTc >450ms for women or >430 msec for men, or 1st degree or higher conduction block.
5. History of unexplained syncope or cardiac syncope.
6. Serum AST and ALT value >2.0 times the upper normal limit.
7. Active infection (acute or chronic).
8. History of diabetes.
9. History of macular edema or uveitis.
10. History of lymphopenia.
11. History of acquired or inherited immune deficiency syndrome, including leukopenia.
12. History of severe untreated chronic obstructive sleep apnea.
13. Exposure to any other agent currently under investigation for the treatment of patients with ALS (off-label use or investigational) within 30 days of the Baseline Visit.
14. Presence of tracheostomy.
15. Use of non-invasive ventilation for hypoventilation due to ALS (such as BiPAP).
16. Presence of feeding tube.
17. Presence of diaphragmatic pacing system.
18. The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, according to PI judgment, or a history of active substance abuse within the prior year.
19. Clinically significant history of unstable or severe cardiac, oncologic, hepatic, or renal disease, or other medically significant illness.
20. Pregnant women or women currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Berry, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - University of California, Irvine, Orange, California
  - Georgia Regents University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Methodist Neurological Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ALS Therapy Development Institute (ALS TDI) — http://www.als.net
- See also: Northeast ALS Consortium (NEALS) — http://www.alsconsortium.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gilenya (Fingolimod) | Placebo
Started | 18 | 10
Randomized | 19 | 11
Completed | 16 | 10
Not Completed | 2 | 0
Not completed — Discontinued Study Drug | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gilenya (Fingolimod) | Placebo | Total
Number analyzed (Participants) | 18 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (8.0) | 55.1 (11.3) | 55.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 17 | 9 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 18 | 8 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 10 | 28
Months Since Symptom Onset [Mean (Standard Deviation); unit: Months] | 12.6 (4.8) | 15.0 (6.2) | 13.5 (5.3)
Months Since Diagnosis [Mean (Standard Deviation); unit: Months] | 5.5 (3.9) | 6.0 (4.0) | 5.7 (3.9)
El Escorial Criteria (EEC) [Number; unit: participants] — El Escorial Criteria (EEC) lists out the criteria for the diagnosis of Amyotrophic Lateral Sclerosis utilizing clinical, electrophysiological or neuropathic examinations.
  participants
    Definite | 11 | 4 | 15
    Probable | 6 | 3 | 9
    Probable Laboratory Supported | 1 | 3 | 4
Bulbar Onset [Number; unit: participants]
  Bulbar Onset | 2 | 4 | 6
  Other | 16 | 6 | 22
Riluzole Usage at Screening [Number; unit: participants]
  On riluzole at screening | 11 | 6 | 17
  Not on riluzole at screening | 7 | 4 | 11
Forced Expiratory Volume (FEV1) (max %-predicted) [Mean (Standard Deviation); unit: % of Predicted Max Value] — Forced Expiratory Volume (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. It will be measured using procedures analogous to those described for the upright SVC.
  % of Predicted Max Value | 83.5 (16.1) | 81.4 (27.9) | 82.8 (20.6)
ALS Functional Rating Scale - Revised (ALSFRS-R) Total Score [Mean (Standard Deviation); unit: Score on a Scale] — The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.
  Score on a Scale | 38.8 (4.1) | 37.9 (5.8) | 38.5 (4.7)
Slow Vital Capacity (max %-predicted) [Mean (Standard Deviation); unit: % of Predicted Max Value] — The vital capacity (VC) (percent of predicted normal) was determined using the slow VC method. Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation. A subject's VC depends on their age, sex and height. The value is recorded as a percent of predicted normal.
  % of Predicted Max Value | 92.8 (18.5) | 82.8 (21.9) | 89.2 (20.0)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meter^2 (kg/m^2)] | 26.1 (3.0) | 26.3 (4.9) | 26.2 (3.7)

OUTCOME MEASURES:

1. Secondary Outcome: Lymphocyte (T-Cell) Subset Trajectories
Description: Gilenya (fingolimod) has been shown to successfully reduce circulating lymphocytes (a type of white blood cell) by blocking their egress (exit) from the lymph nodes. A secondary objective of the study is to quantify the effect of the treatment on circulating lymphocyte populations in patients with ALS.
Time Frame: Week 0, Week 2, and Week 4
Measure: Mean (95% Confidence Interval); unit: 10^3/uL
Arm/Group | Gilenya (Fingolimod) | Placebo
Number analyzed (Participants) | 18 | 10
10^3/uL
  Week 0 | 1.751 [1.527 to 2.008] | 1.751 [1.572 to 2.008]
  Week 2 | 0.580 [0.491 to 0.685] | 1.732 [1.402 to 2.140]
  Week 4 | 0.499 [0.399 to 0.623] | 1.822 [1.357 to 2.447]
Statistical Analysis 1: Comparison: Gilenya (Fingolimod) vs Placebo; Fingolimod vs. Placebo Weeks 0-4; Test type: Superiority or Other; p = 0.746, Random slopes model; Slope = 1.40, 95% CI 2-sided [-7.17 to 9.96], Standard Error of Mean 4.30

2. Primary Outcome: ALSFRS-R Total Score at Weeks 0, 2, 4 and 8
Description: The ALSFRS-R is a quickly administered (5 minutes) ordinal rating scale (ratings 0-4) used to determine subjects' assessment of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS. Initial validity was established by documenting that in ALS patients, change in ALSFRS-R scores correlated with change in strength over time, was closely associated with quality of life measures, and predicted survival.
Time Frame: Week 0, Week 2, Week 4 and Week 8
Population: The reported results are model estimates from a model that estimates a single baseline value across all randomized participants, i.e., reflecting the true state of the population prior to randomization.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Gilenya (Fingolimod) | Placebo
Number analyzed (Participants) | 18 | 10
scores on a scale
  Week 0 | 38.60 [36.4 to 40.8] | 38.60 [36.4 to 40.8]
  Week 2 | 38.15 [35.8 to 40.5] | 38.29 [35.8 to 40.8]
  Week 4 | 38.03 [35.6 to 40.5] | 37.88 [35.3 to 40.5]
  Week 8 | 36.74 [34.1 to 39.4] | 37.10 [34.2 to 40.0]
Statistical Analysis 1: Comparison: Gilenya (Fingolimod) vs Placebo; Fingolimod vs. Placebo Weeks 0-4; Test type: Superiority or Other; p = 0.780, Random slopes model; Slope = 0.25, 95% CI 2-sided [-1.53 to 2.03], Standard Error of Mean 0.89

3. Primary Outcome: Change in Slow Vital Capacity Score (SVC)
Description: The vital capacity (VC) (percent of predicted normal) was determined using the slow VC method. Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation. A subject's VC depends on their age, sex and height. The value is recorded as a percent of predicted normal.
Time Frame: Week 0, Week 2, Week 4 and Week 8
Measure: Mean (95% Confidence Interval); unit: Percentage of predicted max value
Arm/Group | Gilenya (Fingolimod) | Placebo
Number analyzed (Participants) | 18 | 10
Percentage of predicted max value
  Week 0 | 88.28 [84.9 to 91.7] | 88.28 [84.9 to 91.7]
  Week 2 | 88.54 [85.8 to 91.3] | 88.54 [85.8 to 91.3]
  Week 4 | 86.51 [83.4 to 89.6] | 86.70 [82.6 to 90.8]
  Week 8 | 86.02 [83.1 to 89.0] | 87.59 [83.4 to 91.8]
Statistical Analysis 1: Comparison: Gilenya (Fingolimod) vs Placebo; Fingolimod vs. Placebo Weeks 0-4; Test type: Superiority or Other; p = 0.823, Random slopes model; Slope = -0.51, 95% CI 2-sided [-5.00 to 3.99], Standard Error of Mean 2.26

4. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced Expiratory Volume (FEV1): Forced Expiratory Volume (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Screening, Week 0, Week 2, and Week 4
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage of predicted max value
Arm/Group | Gilenya (Fingolimod) | Placebo
Number analyzed (Participants) | 18 | 10
Percentage of predicted max value
  Screening | 84.70 [78.7 to 90.7] | 84.70 [78.7 to 90.7]
  Week 0 | 81.93 [76.3 to 87.5] | 81.93 [76.3 to 87.5]
  Week 2 | 81.19 [74.8 to 87.5] | 80.30 [72.9 to 87.7]
  Week 4 | 80.38 [73.3 to 87.5] | 78.16 [69.5 to 86.8]

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) / Slow Vital Capacity (SVC) Ratio
Description: Forced Expiratory Volume (FEV1): Forced Expiratory Volume (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
  Slow Vital Capacity (SVC): Vital Capacity is the maximum amount of air a person can expel from the lungs after a maximum inhalation. A subject's VC depends on their age, sex and height. The value is recorded as a percent of predicted normal.
Time Frame: Screening, Week 0, Week 2, and Week 4
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage of predicted max value
Arm/Group | Gilenya (Fingolimod) | Placebo
Number analyzed (Participants) | 18 | 10
Percentage of predicted max value
  Screening | 77.39 [70.0 to 84.8] | 77.39 [70.0 to 84.4]
  Week 0 | 74.36 [67.9 to 80.8] | 74.36 [67.9 to 80.8]
  Week 2 | 75.46 [69.0 to 81.9] | 73.14 [65.7 to 80.6]
  Week 4 | 76.34 [69.7 to 83.0] | 71.49 [63.3 to 79.7]
Statistical Analysis 1: Comparison: Gilenya (Fingolimod) vs Placebo; Fingolimod vs. Placebo Weeks 0-4; Test type: Superiority or Other; p = 0.294, Random slopes model; Slope = 4.27, 95% CI 2-sided [-3.78 to 12.33], Standard Error of Mean 4.04

ADVERSE EVENTS:
Arm/Group | Gilenya (Fingolimod) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/10
Other Adverse Events (participants affected / at risk) | 15/18 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gilenya (Fingolimod) (N=18) | Placebo (N=10)
Blood pressure increase (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Electrocardiogram QT prolonged (Cardiac disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 3 (3)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes